CLINICAL TRIAL: NCT01074580
Title: High Frequency Ultrasound and Contrast Enhanced Ultrasound of Patients Treated for Deterioration of Crohn's Disease
Brief Title: Contrast Enhanced Ultrasonography (CEUS) of Patients With Crohn's Disease
Status: Terminated | Type: Observational
Why Stopped: Did not get enough patients
Sponsor: Haukeland University Hospital (Other)
Collaborators: University of Bergen (Other); Abbott (Industry)
Responsible Party: Sponsor
Other Study IDs: 22209
Record Dates: First submitted 2010-02-23; First posted 2010-02-24 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Crohn's Disease
Keywords: Crohn's disease; sonography; contrast enhanced ultrasound
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Mucosal biopsies from the colon and terminal ileum.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Deterioration, Crohn's disease: Patients > 18 years old with a deterioration of Crohn's disease defined by CDAI >150 and requiring treatment with systemic steroids or TNF alfa inhibitors

SUMMARY:
The purpose of this study is investigate if high frequency sonography and contrast enhanced sonography can be used to predict remission in patients with deterioration of Crohn's disease treated with steroids or tumor necrosis factor (TNF) alfa inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Deterioration of Crohn's disease
* CDAI>150
* Treated with systemic steroids or TNF alfa inhibitors
* Lesion found on ultrasound

Exclusion Criteria:

* Disease location not reachable with ileocolonoscopy
* Pregnancy
* Acute coronary disease
* Unstable coronary disease
* Previous allergic reaction to SonoVue or its components

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for deterioration of Crohn's disease either in the out patient clinic or the medical ward of Haukeland University Hospital.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2009-11; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Remission defined by Crohns disease activity index (CDAI)<150 | 52 weeks from inclusion

SECONDARY OUTCOMES:
Surgical treatment for Crohn's disease during follow up. (Surgery for perianal disease not included.) | 52 weeks
Mucosal healing on ileocolonoscopy. Defined by Simple Endoscopic Index for Crohn's disease (SES-CD) | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Trygve Hausken, PhD, Study Director — Nastional Center of Gastroenterological Ultrasonography, Haukeland University Hospital, Bergen, Norway
Locations (1):
- Department of Medicine, Haukeland University Hospital, Bergen, Hordaland, Norway